CLINICAL TRIAL: NCT00816478
Title: Effect of Galactose on Permeability Factor in Patients With Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: Effect of Oral Galactose on Focal Segmental Glomerulosclerosis (FSGS) Permeability Factor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed by Institutional Review Board
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Howard Trachtman MD, principal investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEPHCURE 1
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: FSGS; Permeability factor; Galactose; Primary FSGS, resistant to immunosuppressive medication
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Galactose
  Interventions: Drug: Galactose

INTERVENTIONS:
Drug: Galactose — Oral galactose, 0.2 g/kg/dose twice daily for 28 days

SUMMARY:
This study is a proof-of-concept clinical study designed to test the hypothesis that oral administration of galactose can lower the level of a circulating factor that increases glomerular permeability to albumin in patients with resistant FSGS.

DETAILED DESCRIPTION:
Patients with resistant FSGS have persistent proteinuria and a high risk of progression to end stage kidney disease (ESKD). A circulating factor that increases glomerular permeability to albumin (Palb) has been detected in over 50% of these patients. While the molecular identity of the factor has not been fully established, in vitro studies and limited clinical experience suggest that galactose can reduce the level of the FSGS permeability factor.

This study is a pilot study to determine if oral administration of galactose can lower the circulating level of the FSGS permeability factor.

Two groups of patients with biopsy proven primary FSGS who are resistant to steroids and one other immunosuppressive agents will be studied:

l. FSGS, pre-ESKD 2. FSGS, with ESKD on renal replacement therapy

The only eligibility factor is presence of the FSGS permeability factor.

Five patients will be included in each group.

The experimental intervention is administration of galactose, orally, 0.2 g/kg body weight/dose twice daily. the duration of treatment will be 28 days,.

Patients will be seen on days 0, 14, and 28 of treatment. They will be seen at week 8, 16 and 24 after discontinuation of the galactose.

Physical examination and routine laboratory tests (SMAC, CBC, urine protein:creatinine ratio in an early morning sample) will be done at each visit. The FSGS permeability factor will be assayed at days 0 and 28 of treatment and 6 months after discontinuation of the galactose. The permeability factor will be tested in the laboratory of Virginia Savin MD (Medical college of Wisconsin) using previously described methods.

All other treatments will be unchanged during the 28 day oral galactose Treatment Period.

The study will be analyzed based on the number of patients in whom the FSGS permeability factor is lowered to normal levels.

ELIGIBILITY:
Inclusion Criteria:

* Primary FSGS
* Resistance to steroids and another immunosuppressive medication

Exclusion Criteria:

* Secondary FSGS

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Reduction in FSGS permeability factor | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, MD, Principal Investigator — Schneider Children's Hospital

REFERENCES:
- [Background] Trachtman H, Greenbaum LA, McCarthy ET, Sharma M, Gauthier BG, Frank R, Warady B, Savin VJ. Glomerular permeability activity: prevalence and prognostic value in pediatric patients with idiopathic nephrotic syndrome. Am J Kidney Dis. 2004 Oct;44(4):604-10. PMID 15384010